CLINICAL TRIAL: NCT06518213
Title: Efficacy and Safety of First-line Antiretroviral Therapy (ART) With Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) Introduced at the First Clinical Visit: a Real-life Retrospective Single Arm Single Center Study
Brief Title: Efficacy and Safety of First-line ART With BIC/FTC/TAF Introduced at the First Clinical Visit
Status: Completed | Type: Observational
Sponsor: University Hospital for Infectious Diseases, Croatia (Other)
Responsible Party: Sponsor
Other Study IDs: UHID-09
Record Dates: First submitted 2024-07-12; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections
Keywords: HIV; bictegravir; rapid start; same-day initiation
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Cohort receiving BIC/FTC/TAF as a rapid start, same-day initiation ART: All included subjects (one group, no control group) were started therapy with BIC/FTC/TAF (co-formulated in one tablet of Biktarvy® consisting of 50 mg of bictegravir, 200 mg of emtricitabine and 25 mg of tenofovir alafenamide) within 24 hours of inclusion in care and continued for 12 months.

SUMMARY:
Bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF) is a recommended first-line antiretroviral regimen. Croatia has a centralized care for people living with HIV (PLWH) and all persons are seen and treated in a single center, preferably in a same-day initiation model whenever suitable. This retrospective cohort study evaluated antiretroviral therapy (ART) naïve PLWH who initiated BIC/FTC/TAF, in a same-day model. The goal of the study is to assess safety and efficacy of this model by collecting information from the electronic database of the Croatian HIV Reference Centre.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositivity confirmed by a fourth generation test
* the subject had not previously taken ART
* ART was started within 24 hours of the first examination

Exclusion Criteria:

* persons under 18 years of age
* people who are pregnant, breastfeeding or planning to become pregnant
* unacceptable interaction with a drug that the subject is already taking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In Croatia, all people living with HIV are treated at the University Hospital for Infectious Diseases (UHID) in Zagreb in the HIV Outpatient Department. Included in the study were all patients who entered HIV care in the period from May 2019 to December 2022 and met the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Virological suppression (HIV-1 RNA below 50 copies/mL plasma) | 12±3 months of ART (BIC/FTC/TAF)
  Virological suppression (HIV-1 RNA below 50 copies/mL plasma) after 12±3 months of antiretroviral treatment with first-line ART (BIC/FTC/TAF) initiated at first clinical contact

SECONDARY OUTCOMES:
HIV-1 RNA 50-200 copies/mL | 6 and 12 months of treatment
  HIV-1 RNA 50-200 copies/mL of plasma after 6 and 12 months of treatment
HIV-1 RNA above 200 copies/mL | 6 and 12 months of treatment
  HIV-1 RNA above 200 copies/mL of plasma after 6 and 12 months of treatment
Virological failure | 6 and 12 months of treatment
  Virological failure (HIV-1 RNA above 50 copies/mL) after 6 and 12 months of treatment with BIC/FTC/TAF
Number of CD4+ T-lymphocytes | 6 and 12 months of treatment
  Change in the number of CD4+ T-lymphocytes per microL of blood compared to the initial value after 6 and 12 months of treatment
Change in CD4+/CD8+ T-lymphocytes ratio | 6 and 12 months of treatment
  Change in ratio of CD4+ and CD8+ T-lymphocytes measured after 6 and 12 months of treatment
Side effect to the drug BIC/FTC/TAF | through study completion, an average of 1 year
  Side effect to the administered medication which required discontinuation of treatment
Change in weight | 6 and 12 months of treatment
  Change in patient's weight in kilograms measured after 6 and 12 months of treatment
Change in eGFR | 6 and 12 months of treatment
  Change in estimated glomerular filtration rate (mL/min/1.73 m2) measured after 6 and 12 months of treatment
Change in liver enzymes | 6 and 12 months of treatment
  Change in liver enzymes aspartate aminotransferase (AST), alanine aminotransferase (ALT) and gamma-glutamyl transpeptidase (GGT) concentration (U/L) measured after 6 and 12 months of treatment
Lipids concentration | 6 and 12 months of treatment
  Change in lipids (total cholesterol, LDL, HDL and triglycerides) concentration (mmol/L) measured after 6 and 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Josip Begovac, Prof., Principal Investigator — University Hospital for Infectious Diseases ''Dr. Fran Mihaljevic''
Locations (1):
- University Hospital for Infectious Diseases ''Dr. Fran Mihaljevic'', Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bogdanic N, Bendig L, Lukas D, Zekan S, Begovac J. Timeliness of antiretroviral therapy initiation in the era before universal treatment. Sci Rep. 2021 May 18;11(1):10508. doi: 10.1038/s41598-021-90043-7. PMID 34006927
- [Result] Mounzer K, Brunet L, Fusco JS, Mcnicholl IR, Diaz Cuervo H, Sension M, Mccurdy L, Fusco GP. Advanced HIV Infection in Treatment-Naive Individuals: Effectiveness and Persistence of Recommended 3-Drug Regimens. Open Forum Infect Dis. 2022 Jan 13;9(3):ofac018. doi: 10.1093/ofid/ofac018. eCollection 2022 Mar. PMID 35169590
- [Result] Camici M, Gagliardini R, Lanini S, Del Duca G, Mondi A, Ottou S, Plazzi MM, De Zottis F, Pinnetti C, Vergori A, Grilli E, Mastrorosa I, Mazzotta V, Paulicelli J, Bellagamba R, Cimini E, Tartaglia E, Notari S, Tempestilli M, Cicalini S, Amendola A, Abbate I, Forbici F, Fabeni L, Girardi E, Vaia F, Maggi F, Antinori A. Rapid ART initiation with bictegravir/emtricitabine/tenofovir alafenamide in individuals presenting with advanced HIV disease (Rainbow study). Int J Antimicrob Agents. 2024 Jan;63(1):107049. doi: 10.1016/j.ijantimicag.2023.107049. Epub 2023 Dec 5. PMID 38056572
- [Result] Bachelard A, Isernia V, Charpentier C, Benalycherif A, Mora M, Donadille C, Duvivier C, Lacombe K, El Mouhebb M, Spire B, Landman R, Descamps D, Peytavin G, Assoumou L, Ghosn J; FAST study group. Same-day initiation of bictegravir/emtricitabine/tenofovir alafenamide: Week 48 results of the FAST study-IMEA 055. J Antimicrob Chemother. 2023 Mar 2;78(3):769-778. doi: 10.1093/jac/dkad008. PMID 36659824
- [Result] Hidalgo-Tenorio C, Sequera S, Vivancos MJ, Vinuesa D, Collado A, Santos IL, Sorni P, Cabello-Clotet N, Montero M, Font CR, Terron A, Galindo MJ, Martinez O, Ryan P, Omar-Mohamed M, Albendin-Iglesias H, Javier R, Ruz MAL, Romero A, Garcia-Vallecillos C. Bictegravir/emtricitabine/tenofovir alafenamide as first-line treatment in naive HIV patients in a rapid-initiation model of care: BIC-NOW clinical trial. Int J Antimicrob Agents. 2024 Jun;63(6):107164. doi: 10.1016/j.ijantimicag.2024.107164. Epub 2024 Apr 2. PMID 38574873
- [Result] Ambrosioni J, Rojas Lievano J, Berrocal L, Inciarte A, de la Mora L, Gonzalez-Cordon A, Martinez-Rebollar M, Laguno M, Torres B, Ugarte A, Chivite I, Leal L, de Lazzari E, Miro JM, Blanco JL, Martinez E, Mallolas J. Real-life experience with bictegravir/emtricitabine/tenofovir alafenamide in a large reference clinical centre. J Antimicrob Chemother. 2022 Mar 31;77(4):1133-1139. doi: 10.1093/jac/dkab481. PMID 35040990
- See also: European AIDS Clinical Society guidelines for the management of people living with HIV in Europe — https://www.eacsociety.org/guidelines/eacs-guidelines